CLINICAL TRIAL: NCT07128992
Title: The Impact of Need-driven Treatment of Insulin-Deficient Diabetes on the Care Events, Glycemic Control, Risk Factors, and Complications in the Pirkanmaa Wellbeing Services County, Finland
Brief Title: Need-driven Treatment of the Patients With Type 1 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Saara Metso, Head of the unit of endocrinology, Associate professor, Tampere University Hospital
Other Study IDs: R25006L; T67674 (Other Grant/Funding Number: State funding for university-level health research)
Record Dates: First submitted 2025-06-27; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes (T1D); Glucose Control
Keywords: type 1 diabetes; complication; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults (≥18 years) with type1 diabetes under the care of the Pirkanmaa Wellbeing Service: Eligible participants are patients with type 1 diabetes who use continuous glucose monitoring systems, have no complications or other conditions requiring frequent hospital or outpatient care, and are in good glycemic control (HbA1c < 53 mmol/mol, TIR > 70%, TBR < 4%, TAR > 25%).
  Interventions: Other: Control visit interval

INTERVENTIONS:
Other: Control visit interval — Study investigates whether it is safe to extend the interval of routine calendar-based follow-up visits from every 12 to every 24 months in patients with type 1 diabetes.

SUMMARY:
This prospective study evaluates the safety of extending the interval of routine calendar-based follow-up visits from every 12 months to every 24 months in patients with type 1 diabetes who are in good glycemic control and suitable for remote monitoring. The primary outcome is the proportion of patients who maintain good glycemic control during the 24-month follow-up period.

Participants will attend two in-person visits at baseline (month 0) and at the end of follow-up (month 24), which include a comprehensive clinical examination, assessment of glucose control, and laboratory testing. One remote contact will occur at month 12 for prescription renewal and review of glucose data. Patients may contact their care unit as needed throughout the study. At the baseline and final visits, participants will complete a questionnaire assessing their perceived ability to manage self-care, the safety of the care plan, and their ability to contact their care provider when necessary.

DETAILED DESCRIPTION:
The primary outcome of this study is the proportion of patients who maintain good glycemic control during the 24-month follow-up period. A clinically significant result is defined as no more than 14% of patients (95% confidence interval: 8%-20%) experiencing deterioration in glucose control, indicated by Time in Range (TIR) < 70% or HbA1c > 53 mmol/mol. If at least 125 patients are enrolled, need-based care can be demonstrated to be safe.

The study also evaluates the performance and safety of the "MD Diabetes Huolijono" software application, which issues alerts to healthcare professionals if glucose control worsens or if the patient is hospitalized. Between visits, patients using a Libre sensor with multiple daily insulin injections will be monitored using the MD Diabetes Huolijono system, while other patients will continue standard self-monitoring.

Healthcare contact data will be retrieved from the data service for each participant for the 24 months prior to study enrollment and throughout the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of type 1 diabetes
* Treatment with multiple daily injections or insulin pump therapy
* Duration of diabetes ≥ 1 year
* Good glycemic control over the previous two weeks, defined as:
* HbA1c < 53 mmol/mol
* Time in Range (TIR) > 70%
* Time Below Range (TBR) < 4%
* Time Above Range (TAR) < 25%
* Use of a continuous glucose monitoring system connected via a smartphone application
* Under specialist diabetes care within the Pirkanmaa Wellbeing Services County (Pirha)
* Willing to accept remote diabetes care by granting the diabetes team at Tampere University Hospital access to glucose data
* No need for regular specialist care due to other medical conditions
* Provides informed consent to participate in the study

Exclusion Criteria:

* Age < 18 years
* Duration of diabetes < 1 year
* Pregnancy
* Not using multiple daily injections or insulin pump therapy
* Not using a continuous glucose monitoring system
* Does not accept remote care
* History of diabetic ketoacidosis or severe hypoglycemia within the past 12 months
* Presence of retinopathy
* No retinal imaging performed within the past 12 months
* Urine albumin-creatinine ratio (uACR) > 3 mg/mmol or estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m² on two occasions over a period of more than 3 months
* Undergoing dialysis or post-kidney transplantation
* Cardiovascular disease (excluding hypertension)
* Neuropathy, foot ulcer, or amputation (foot risk category 1-3)
* Scheduled hospital outpatient visits for other specialties within the next 12 months
* Not under specialist diabetes care within the Pirkanmaa Wellbeing Services County (Pirha)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults (≥18 years) with type 1 diabetes in good glucose control and under the care of the Pirkanmaa Wellbeing Services County (Pirha).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in good glycemic control | At the baseline and at 24 months of follow-up
  Percentage of patients with TIR > 70%, GMI < 53 mmol/mol, and HbA1c < 53 mmol/mol

CONTACTS AND LOCATIONS:
Overall Officials: Saara Metso, MD, PhD, Principal Investigator — Tampere University Hospital, Pirkanmaa Wellbeing County

IPD SHARING:
Plan to Share IPD: Undecided